CLINICAL TRIAL: NCT07017764
Title: Combined Effect of Core Stability and Theraband Resisted Exercises on Gait Parameters in Lower Limb Burn
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noura Mohamed Fouad Hussein, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005543
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Core stability exercises + Theraband resisted exercises + Traditional physical therapy program (Experimental): This group will be composed of 22 patients with second degree lower limb burn of thermal injury. Patients will receive core stability and theraband resisted exercises in addition to a traditional physical therapy program in the form of ambulation, stretching exercises for the muscles of the lower limbs and range of motion exercises. Exercises will be applied for 3 times a week for 8 consecutive weeks.
  Interventions: Other: Core stability exercises; Other: Theraband resisted exercises; Other: Traditional physical therapy program
- Core stability exercises + Traditional physical therapy program (Active Comparator): This group will be composed of 22 patients with second degree lower limb burn of thermal injury. Patients will receive core stability exercises in addition to traditional physical therapy program in the form of ambulation, stretching exercises for the muscles of the lower limbs and range of motion exercises.
  Exercises will be applied for 3 times a week for 8 consecutive weeks.
  Interventions: Other: Core stability exercises; Other: Traditional physical therapy program
- Theraband resisted exercises + Traditional physical therapy program (Active Comparator): This group will be composed of 22 patients with second degree lower limb burn of thermal injury. Patients will receive theraband resisted exercises in addition to traditional physical therapy program in the form of ambulation, stretching exercises for the muscles of the lower limbs and range of motion exercises. Exercises will be applied for 3 times a week for 8 consecutive weeks.
  Interventions: Other: Theraband resisted exercises; Other: Traditional physical therapy program

INTERVENTIONS:
Other: Core stability exercises — Core stability exercises will be performed for 8 weeks, 3 times per week, 30 minutes per session. The program includes bed, wedge, and Swiss ball exercises. Bed exercises involve bridges, curl-ups, bird dog, and side bridges. Wedge exercises include curl-ups in various arm positions. Ball exercises involve bridges, curl-ups, bird dog, and push-ups. Each position is held for 7 seconds with 10 seconds of rest, repeated 10 times per set, for 2 sets per session with 60 seconds rest between sets.
  Arms: Core stability exercises + Theraband resisted exercises + Traditional physical therapy program; Core stability exercises + Traditional physical therapy program
Other: Theraband resisted exercises — TheraBand resisted exercises will be performed for 8 weeks, 3 times per week, 30 minutes per session. Each session includes a 5-minute warm-up (stretching and joint mobilization), 30 minutes of resistance training for lower limbs (ankle, knee, hip), and a 5-minute cool-down with deep breathing and self-massage. Exercises include ankle flexion/extension, knee flexion/extension, and hip flexion/extension, abduction/adduction using elastic bands. Movements are done alternately on both sides, 10 reps each, 3 sets per session, with 1-2 min rest between sets. Yellow bands are used in weeks 1-4; green bands in weeks 5-8.
  Arms: Core stability exercises + Theraband resisted exercises + Traditional physical therapy program; Theraband resisted exercises + Traditional physical therapy program
Other: Traditional physical therapy program — All patients will receive a traditional physical therapy program consisting of ambulation training, stretching exercises for lower limb muscles, and range of motion exercises.

SUMMARY:
The purpose of the study is designed to evaluate the combined effect of core stability and theraband resisted exercises on gait parameters in lower limb burn.

DETAILED DESCRIPTION:
Impairments such as pain and decreased range of motion (ROM) may develop in patients who have thermal burn on their lower extremities. These impairments may contribute to an individual's functional limitations, including impaired gait. For example, patients with burns on planter aspects of their feet have difficulty with ambulation because of pain. Also, individuals with burns on Achilles tendon area or popliteal space have difficulty with ambulation because of decreased ROM of the ankle and knee, respectively. Burns on the lower extremities may cause changes in step length and deviations in heel-toe gait pattern as the patient tries to avoid bearing down on the affected extremity. Patients with lower extremity burns may walk with decreased stance phase on the affected lower extremity, a decreased swing phase on the unaffected lower extremity, and a wider base of support.

One goal of core stability is to optimize motor control of the lumbo-pelvic region to sustain functional stability in neutral positions and contribute to producing and transmitting energy from the trunk to the limbs.

Core stability aims to provide proximal stability to facilitate distal mobility and power generation, particularly in movements in which the stability of the spine is involved.

Since 1980 and with resounding research and outcomes, the use of the Theraband as an elastic resistance training (ERT) modality has become a common treatment intervention. Improved functional ability, enhanced strength and endurance with higher muscular activation, and reduced injury risks are some of its advantages.

Systematic resistance exercise, results in gait analysis changes in the synergy ratios of different muscle groups, while resistance training using elastic bands increases muscle strength levels and improves explosive strength. Also, evident is the effect of elastic resistance exercise in increasing the range of motion, the flexibility of movement, walking ability (effect on kinematic parameters in gait analysis) and the promotion of various skills of everyday life. Furthermore, the need for this study is developed from the lack of information in the published studies about the effect of core stability and theraband resisted exercises on gait parameters in lower limb burn. So, this study is designed to evaluate the combined effect of core stability and theraband resisted exercises on gait parameters in lower limb burn.

ELIGIBILITY:
Inclusion Criteria:

* Patients will suffer from second degree lower limb burn (Partial thickness of thermal injury).
* Total body surface area (TBSA) for the burns will be ranged from 20% to 25% .
* Patients will begin the training program after complete skin closure from (1-2) weeks.
* All patients enrolled to the study will have their informed consent.

Exclusion Criteria:

* Patients who had an open wound at or near treatment site.
* Patients who had chemical or electrical burn.
* Neurological and renal disorders.
* Malignant conditions.
* Psychiatric illness, severe behavior or cognitive disorders.
* Use of neurological drugs that influence gait parameters.
* History of lower extremity injuries with in the last 6 months.
* History of muscular/ neural aliments (myopathy, myositis, peripheral neuropathy, muscular dystrophy).
* Postural abnormality in the upper or lower extremities (such as kyphosis, lordosis, forward head, knee valgus and knee varus).
* Surgery or fracture within a year before the study.
* Insulin-dependent diabetes.
* Joint rheumatoid arthritis.
* Diagnosed cerebrovascular disease or any other disease that interferes with sensory input.
* Lower extremity rotational deformities (increased anteversion, tibial torsion or pes planovalgus).
* Hormonal changes.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-06-11 (Estimated); Primary Completion 2025-10-11 (Estimated); Study Completion 2025-10-26 (Estimated)

PRIMARY OUTCOMES:
Step length | 8 weeks
  Using two-dimentional (2D) videobased gait assessment system, the distance between the ipsilateral and contralateral heel strikes will be measured in meters before and after treatment for all participants in the three groups.
Stride length | 8 weeks
  Using two-dimentional (2D) videobased gait assessment system, the distance between two consecutive heel strikes of the same foot will be measured in meters before and after treatment for all participants in the three groups.
Step width | 8 weeks
  Using two-dimentional (2D) videobased gait assessment system, the distance between the centre lines of the two feet, perpendicular to the plane of walking will be measured in centimeters before and after treatment for all participants in the three groups.
Step time | 8 weeks
  Using two-dimentional (2D) videobased gait assessment system, the time between ipsilateral and contralateral heel strikes will be measured in seconds before and after treatment for all participants in the three groups.
Stride time | 8 weeks
  Using two-dimentional (2D) videobased gait assessment system, the time elapsed between the first contact of two consecutive footsteps of the same foot will be measured in seconds before and after treatment for all participants in the three groups.
Cadence | 8 weeks
  Using two-dimentional (2D) videobased gait assessment system, the number of steps in a minute, [steps/ minute]. It will be measured in seconds before and after treatment for all participants in the three groups.
Velocity | 8 weeks
  Using two-dimentional (2D) videobased gait assessment system, the distance covered by the body in unit time, (meter/minute) = Step length × Cadence. It will be measured in seconds before and after treatment for all participants in the three groups.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Mohamed Othman, PhD, Study Chair — Professor, Cairo university; Tarek Ahmed Amer, PhD, Study Director — Professor, Cairo university; Noha Mohamed Kamel, PhD, Study Director — Lecturer, Cairo university
Locations (1):
- El Mahalla General Hospital and Burn Center in Mansoura University Hospital, Al Mansurah, Egypt